CLINICAL TRIAL: NCT06174298
Title: The Role of Granulocyte Colony Stimulating Factor in Embryo Transfer Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Newlife Fertility Centre (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFC-2023-001
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Infertility; Infertility,Female; Infertility; Female, Nonimplantation; Infertility Unexplained; Infertility of Uterine Origin
Keywords: Infertility; Embryo Transfer; GCSF; Granulocyte Colony-Stimulating Factor; Filgrastim; Neupogen; Implantation
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GCSF-Supplemented Embryo Transfer Media (Experimental): Intervention Group Frozen Embryo Transfers: Cryopreserved embryos will be thawed according to the Kitazato thawing protocol and will be subsequently transferred to a center-well dish containing 1 mL of embryo transfer media supplemented with GCSF. The embryos will be cultured in this medium for approximately 3 hours before the embryo transfer (ET) procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Fresh Embryo Transfers: On day 5 or 6 of culture, viable embryos will be transferred into a center-well dish containing 1 mL of embryo transfer media supplemented with GCSF. The embryos will be cultured in this medium for approximately 3 hours before the ET procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor (Filgrastim)
- Standard Embryo Transfer Media (Placebo Comparator): Control Group Fresh Embryo Transfers: On day 5 or 6 of culture, viable embryos will be transferred into a center-well dish containing 1 mL of standard embryo transfer media. The embryos will be cultured in this medium for approximately 3 hours before the embryo transfer (ET) procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Control Group Frozen Embryo Transfers: Cryopreserved embryos will be thawed according to the Kitazato thawing protocol and will be subsequently transferred to a center-well dish containing 1 mL of standard embryo transfer media. The embryos will be cultured in this medium for approximately 3 hours before the ET procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Interventions: Other: Standard Embryo Transfer Media

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor (Filgrastim) — Intervention Group Fresh Embryo Transfers: On day 5 or 6 of culture, viable embryos will be transferred into a center-well dish containing 1 mL of embryo transfer media supplemented with GCSF. The embryos will be cultured in this medium for approximately 3 hours before the embryo transfer (ET) procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Intervention Group Frozen Embryo Transfers: Cryopreserved embryos will be thawed according to the Kitazato thawing protocol and will be subsequently transferred to a center-well dish containing 1 mL of embryo transfer media supplemented with GCSF. The embryos will be cultured in this medium for approximately 3 hours before the ET procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Other Names: Neupogen; Filgrastim
  Arms: GCSF-Supplemented Embryo Transfer Media
Other: Standard Embryo Transfer Media — Control Group Fresh Embryo Transfers: On day 5 or 6 of culture, viable embryos will be transferred into a center-well dish containing 1 mL of embryo transfer media. The embryos will be cultured in this medium for approximately 3 hours before the embryo transfer (ET) procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Control Group Frozen Embryo Transfers: Cryopreserved embryos will be thawed according to the Kitazato thawing protocol and will be subsequently transferred to a center-well dish containing 1 mL of embryo transfer media. The embryos will be cultured in this medium for approximately 3 hours before the ET procedure. During the ET procedure, the same media will be used to fill the ET syringe and catheter that will be used to deposit the embryos into the uterus by the physician.
  Arms: Standard Embryo Transfer Media

SUMMARY:
The goal of this clinical trial is to test the effect of granulocyte colony-stimulating factor (G-CSF, A.K.A. Filgrastim) in infertility patients undergoing in vitro fertilization (IVF) treatment. The main question it aims to answer is:

Can in vitro fertilization-embryo transfer (IVF-ET) outcomes be improved by supplementing the transfer media with Granulocyte colony-stimulating factor (GCSF)?

Participants will undergo their embryo transfer as per the normal clinic protocol but will be randomized to either receive the standard embryo transfer media or the GCSG-supplemented transfer media.

Researchers will compare the GCSF and standard transfer media groups to see if clinical outcomes are improved (i.e., implantation rate, pregnancy, clinical pregnancy rate, live birth rate).

DETAILED DESCRIPTION:
Please see uploaded study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Recruited subjects will either be undergoing a fresh IVF-ET cycle in which the embryo(s) generated from the initial treatment cycle are transferred during that same cycle (i.e., on day 5 or 6 post-egg retrieval) or an FET cycle in which the embryo(s) transferred were generated in a previous IVF cycle and were cryopreserved for subsequent warming and transfer.

Exclusion Criteria:

* Patients with uterine factor or severe male factor infertility will be excluded.
* Patients who have had previous IVF failures will be excluded.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological Females (cisgender women)
Enrollment: 300 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Implantation Rate | From enrollment to the time of 6-week ultrasound.
  Number of embryos implanted (i.e. number of gestational sacs observed under ultrasound guidance) divided by total number of embryos transferred
Clinical Pregnancy Rate | From enrollment to the time of 6-week ultrasound.
  Number of patients with fetal heartbeats detected at time of 6-week ultrasound divided by the total number of patients in that group.
Pregnancy Rate | From enrollment to the time of blood test at 10 days post-ET.
  Number of patients with a positive beta-human chorionic gonadotropin (bhCG) pregnancy blood test at 10 days post-ET divided by the total number of patients in that group.
Live Birth Rate | From enrollment to the time of birth (up to 9-months post-ET).
  Total Number of infants born divided by the total number of embryo transfers performed (i.e., patients) in that group.

SECONDARY OUTCOMES:
Spontaneous Abortion Rate | From enrollment to the time of pregnancy loss (up to 20 weeks post-ET).
  Number of patients with a confirmed clinical pregnancy who lost their pregnancy before 20 weeks of gestation divided by the total number of patients with confirmed clinical pregnancies.
Biochemical Pregnancy Rate | From enrollment to the time of 6-week ultrasound.
  Number of patients who had a positive beta-human chorionic gonadotropin (bhCG) pregnancy blood test at 10 days post-ET but that did not display a gestational sac/fetal heartbeat at 6-week ultrasound, divided by the total number of patients in that group.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Soliman, M.D., Principal Investigator — Newlife Fertility Centre
Locations (1):
- Newlife Fertility Centre, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolibianakis E, Bourgain C, Albano C, Osmanagaoglu K, Smitz J, Van Steirteghem A, Devroey P. Effect of ovarian stimulation with recombinant follicle-stimulating hormone, gonadotropin releasing hormone antagonists, and human chorionic gonadotropin on endometrial maturation on the day of oocyte pick-up. Fertil Steril. 2002 Nov;78(5):1025-9. doi: 10.1016/s0015-0282(02)03323-x. PMID 12413988
- [Background] Devroey P, Bourgain C, Macklon NS, Fauser BC. Reproductive biology and IVF: ovarian stimulation and endometrial receptivity. Trends Endocrinol Metab. 2004 Mar;15(2):84-90. doi: 10.1016/j.tem.2004.01.009. PMID 15036255
- [Background] Yan J, Wu K, Tang R, Ding L, Chen ZJ. Effect of maternal age on the outcomes of in vitro fertilization and embryo transfer (IVF-ET). Sci China Life Sci. 2012 Aug;55(8):694-8. doi: 10.1007/s11427-012-4357-0. Epub 2012 Aug 30. PMID 22932885
- [Background] Thum MY, Abdalla HI, Taylor D. Relationship between women's age and basal follicle-stimulating hormone levels with aneuploidy risk in in vitro fertilization treatment. Fertil Steril. 2008 Aug;90(2):315-21. doi: 10.1016/j.fertnstert.2007.06.063. Epub 2007 Oct 22. PMID 17953958
- [Background] Seshadri S, Morris G, Serhal P, Saab W. Assisted conception in women of advanced maternal age. Best Pract Res Clin Obstet Gynaecol. 2021 Jan;70:10-20. doi: 10.1016/j.bpobgyn.2020.06.012. Epub 2020 Aug 7. PMID 32921559
- [Background] Tevkin S, Lokshin V, Shishimorova M, Polumiskov V. The frequency of clinical pregnancy and implantation rate after cultivation of embryos in a medium with granulocyte macrophage colony-stimulating factor (GM-CSF) in patients with preceding failed attempts of ART. Gynecol Endocrinol. 2014 Oct;30 Suppl 1:9-12. doi: 10.3109/09513590.2014.945767. PMID 25200819
- [Background] Sjoblom C, Wikland M, Robertson SA. Granulocyte-macrophage colony-stimulating factor promotes human blastocyst development in vitro. Hum Reprod. 1999 Dec;14(12):3069-76. doi: 10.1093/humrep/14.12.3069. PMID 10601098
- [Background] Ziebe S, Loft A, Povlsen BB, Erb K, Agerholm I, Aasted M, Gabrielsen A, Hnida C, Zobel DP, Munding B, Bendz SH, Robertson SA. A randomized clinical trial to evaluate the effect of granulocyte-macrophage colony-stimulating factor (GM-CSF) in embryo culture medium for in vitro fertilization. Fertil Steril. 2013 May;99(6):1600-9. doi: 10.1016/j.fertnstert.2012.12.043. Epub 2013 Feb 4. PMID 23380186
- [Background] Davari-Tanha F, Shahrokh Tehraninejad E, Ghazi M, Shahraki Z. The role of G-CSF in recurrent implantation failure: A randomized double blind placebo control trial. Int J Reprod Biomed. 2016 Dec;14(12):737-742. PMID 28066833
- [Background] Eftekhar M, Miraj S, Farid Mojtahedi M, Neghab N. Efficacy of Intrauterine infusion of granulocyte colony stimulating factor on patients with history of implantation failure: A randomized control trial. Int J Reprod Biomed. 2016 Nov;14(11):687-690. PMID 27981253
- [Background] Obidniak D, Gzgzyan A, Dzhemlikhanova L, Feoktistov A. Effect of colony-stimulating growth factor on outcome of frozen-thawed embryo transfer in patients with repeated implantation failure. Fertility and Sterility. 2016;106(3):e134-e135.
- [Background] Singh R, Singh M, Jindal A, Jindal P. A prospective randomized controlled study (RCT) of Intra-uterine administration of Granulocyte Colony-Stimulating Factor (G-CSF) before embryo-transfer on resistant thin endometrium in IVF cycles. OXFORD UNIV PRESS GREAT CLARENDON ST, OXFORD OX2 6DP, ENGLAND; 2015:280-280.
- [Background] Barad DH, Yu Y, Kushnir VA, Shohat-Tal A, Lazzaroni E, Lee HJ, Gleicher N. A randomized clinical trial of endometrial perfusion with granulocyte colony-stimulating factor in in vitro fertilization cycles: impact on endometrial thickness and clinical pregnancy rates. Fertil Steril. 2014 Mar;101(3):710-5. doi: 10.1016/j.fertnstert.2013.12.016. Epub 2014 Jan 11. PMID 24424357
- [Background] Scarpellini F, Sbracia M. G-CSF treatment improves IVF outcome in women with recurrent implantation failure in IVF. Journal of Reproductive Immunology. 2012;1(94):103.
- [Background] Aleyasin A, Abediasl Z, Nazari A, Sheikh M. Granulocyte colony-stimulating factor in repeated IVF failure, a randomized trial. Reproduction. 2016 Jun;151(6):637-42. doi: 10.1530/REP-16-0046. Epub 2016 Mar 15. PMID 26980809
- [Background] Würfel W. Approaches to a better implantation. J Assist Reprod Genet. 2000;17(8):473.
- [Background] Rahmati M, Petitbarat M, Dubanchet S, Bensussan A, Chaouat G, Ledee N. Granulocyte-Colony Stimulating Factor related pathways tested on an endometrial ex-vivo model. PLoS One. 2014 Oct 2;9(9):e102286. doi: 10.1371/journal.pone.0102286. eCollection 2014. PMID 25275446
- [Background] Cai L, Jeon Y, Yoon JD, Hwang SU, Kim E, Park KM, Kim KJ, Jin MH, Lee E, Kim H, Jeung EB, Hyun SH. The effects of human recombinant granulocyte-colony stimulating factor treatment during in vitro maturation of porcine oocyte on subsequent embryonic development. Theriogenology. 2015 Oct 15;84(7):1075-87. doi: 10.1016/j.theriogenology.2015.06.008. Epub 2015 Jun 19. PMID 26194698
- [Background] Giacomini G, Tabibzadeh SS, Satyaswaroop PG, Bonsi L, Vitale L, Bagnara GP, Strippoli P, Jasonni VM. Epithelial cells are the major source of biologically active granulocyte macrophage colony-stimulating factor in human endometrium. Hum Reprod. 1995 Dec;10(12):3259-63. doi: 10.1093/oxfordjournals.humrep.a135899. PMID 8822455
- [Background] Zhao Y, Rong H, Chegini N. Expression and selective cellular localization of granulocyte-macrophage colony-stimulating factor (GM-CSF) and GM-CSF alpha and beta receptor messenger ribonucleic acid and protein in human ovarian tissue. Biol Reprod. 1995 Oct;53(4):923-30. doi: 10.1095/biolreprod53.4.923. PMID 8547489
- [Background] Davidson LM, Coward K. Molecular mechanisms of membrane interaction at implantation. Birth Defects Res C Embryo Today. 2016 Mar;108(1):19-32. doi: 10.1002/bdrc.21122. Epub 2016 Mar 10. PMID 26969610
- [Background] Nimbkar-Joshi S, Rosario G, Katkam RR, Manjramkar DD, Metkari SM, Puri CP, Sachdeva G. Embryo-induced alterations in the molecular phenotype of primate endometrium. J Reprod Immunol. 2009 Dec;83(1-2):65-71. doi: 10.1016/j.jri.2009.08.011. Epub 2009 Oct 31. PMID 19880195
- [Background] Zhang L, Xu WH, Fu XH, Huang QX, Guo XY, Zhang L, Li SS, Zhu J, Shu J. Therapeutic role of granulocyte colony-stimulating factor (G-CSF) for infertile women under in vitro fertilization and embryo transfer (IVF-ET) treatment: a meta-analysis. Arch Gynecol Obstet. 2018 Nov;298(5):861-871. doi: 10.1007/s00404-018-4892-4. Epub 2018 Sep 15. PMID 30220024